CLINICAL TRIAL: NCT02501109
Title: A Single-dose, Randomized, Three-period, Crossover Comparative Bioavailability Study of a Novel Formulation of Aripiprazole 10 mg Oral Soluble Film vs the Marketed Formulation Abilify® 10 mg Tablet in Healthy Volunteers
Brief Title: Comparative Bioavailability Study of Aripiprazole 10 mg Oral Soluble Film vs Abilify® 10 mg Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CMG Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMG-ARI-140052
Record Dates: First submitted 2015-06-04; First posted 2015-07-17 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; Oral Soluble Film; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Healthy volunteers will receive Aripiprazole Oral Soluble Film(OSF) 10mg orally a single of dose within 28 days with water.
  Interventions: Drug: Aripiprazole
- Group B (Experimental): Healthy volunteers will receive Aripiprazole Oral Soluble Film(OSF) 10mg orally a single of dose within 28 days without water.
  Interventions: Drug: Aripiprazole
- Gruop C (Experimental): Healthy volunteers will receive the reference drug Abilify tab. 10mg orally a single of dose within 28 days with water.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Healthy volunteers will receive Aripiprazole Oral Soluble Fim(OSF) 10mg orally a single of dose within 28 days
  Other Names: Abilify® 10 mg tablet

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Aripiprazole Oral Soluble Film 10 mg (Test) versus Abilify® 10 mg tablet (Reference) in healthy male volunteers

DETAILED DESCRIPTION:
The proposed study is a single centre, bioavailability, open-label, randomized, single-dose, 3-period, 6-sequence, crossover study under fasting conditions. Each volunteer will be given a single dose of the Test formulation in two study periods (with and without water), and a single dose of the Reference formulation (with water) in the other study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, moderate smoker (no more than 9 cigarettes daily) or non-smoker, ≥45 and ≤65 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight 50.0 kg for males and 45.0 kg for females.
2. Healthy as defined by:
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive method throughout the study and for 42 days after the last study drug administration:
4. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to aripiprazole, dimenhydrinate, benztropine, diphenhydramine or other related drugs.
4. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration.
5. Positive pregnancy test at screening.
6. Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
7. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm), decrease in systolic blood pressure of 20 mmHg or higher, or decrease in diastolic blood pressure of 10 mmHg or higher within 2 to 3 minutes after passing from a supine to a standing position, at screening.
8. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
9. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine (PCP), and crack) within 1 year prior to screening.
10. Use of aripiprazole for a medical condition or in the context of another clinical trial within a period of 42 days prior to the first dosing.
11. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
12. Use of medication other than topical products without significant systemic absorption and hormonal contraceptives:

    * prescription medication within 14 days prior to the first dosing;
    * over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    * a depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to the first dosing.
13. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
14. Hemoglobin <128 g/L (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening.
15. Breast-feeding subject.
16. HAM-D-7 scale score above 3 at screening.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The rate extent of absorption of aripiprazole OSF 10mg versus Abilify ® 10mg tablet | Baseline to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Byung Jo Kim, M.D., Study Director — Development Div.

IPD SHARING:
Plan to Share IPD: Yes